CLINICAL TRIAL: NCT01471041
Title: Vital Access Venous Window Needle Guide for Salvage of AV FistulaE (SAVE) Trial
Brief Title: Safety and Efficacy Study of the Venous Window Needle Guide to Access Arteriovenous (AV)Fistulae
Acronym: SAVE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vital Access Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VA 024
Record Dates: First submitted 2011-11-01; First posted 2011-11-11 (Estimated); Results first posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-04

CONDITIONS: End Stage Renal Disease; AV Fistula; Kidney Failure
Keywords: End Stage Renal Disease; Hemodialysis; AV fistula; Kidney failure
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Venous Window Needle Guide (Experimental): Venous Window Needle Guide will be implanted onto deep, un-cannulatable arteriovenous fistula
  Interventions: Device: Venous Window Needle Guide

INTERVENTIONS:
Device: Venous Window Needle Guide — Subcutaneous, extravascular needle guide made of medical-grade titanium
  Other Names: VWNG

SUMMARY:
The SAVE Study will evaluate the safety and efficacy of the Venous Window Needle Guide in achieving access of a deep, un-cannulatable arteriovenous fistula to complete hemodialysis as prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Deep, uncannulatable, upper extremity arteriovenous fistula
* Minimum arteriovenous fistula flow 400 ml/min
* One year life expectancy

Exclusion Criteria:

* Non-transposed basilic or brachial vein arteriovenous fistula
* History of peripheral vascular disease
* History of cardiovascular disease
* History of cerebral vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Crawford, BA, Study Director — Vital Access
Locations (2):
- United States (2):
  - Ladenheim Dialysis Access Centers, Fresno, California
  - University of Oklahoma - Tulsa, Tulsa, Oklahoma

REFERENCES:
- [Derived] Jennings WC, Galt SW, Shenoy S, Wang S, Ladenheim ED, Glickman MH, Kathuria P, Browne BJ. The Venous Window Needle Guide, a hemodialysis cannulation device for salvage of uncannulatable arteriovenous fistulas. J Vasc Surg. 2014 Oct;60(4):1024-32. doi: 10.1016/j.jvs.2014.04.016. Epub 2014 May 13. PMID 24833247

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Venous Window Needle Guide
Started | 54
Completed | 47
Not Completed | 7

BASELINE CHARACTERISTICS:
Population: ESRD patients treated with HD having a deep, uncanulatable AVF
Arm/Group | Venous Window Needle Guide
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 16
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Use of Venous Window Needle Guide to Obtain Arteriovenous Access for Hemodialysis
Description: Successful cannulation of arteriovenous fistula through the VWNG device and successful hemodialysis achieved within 3 months from index procedure.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Venous Window Needle Guide
Number analyzed (Participants) | 51
participants | 49

2. Secondary Outcome: Arteriovenous Fistula Cannulation Complications While Using the Venous Window Needle Guide
Description: Frequency of complications occuring when cannulating the arteriovenous fistula through the Venous Window Needle Guide
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Venous Window Needle Guide
Number analyzed (Participants) | 54
participants | 14

ADVERSE EVENTS:
Time Frame: 6 mths
Arm/Group | Venous Window Needle Guide
Serious Adverse Events (participants affected / at risk) | 8/54
Other Adverse Events (participants affected / at risk) | 44/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venous Window Needle Guide (N=54)
Stenosis at VWING (Blood and lymphatic system disorders) | 3 (3)
Cannulation pain resulting in VWING removal (Blood and lymphatic system disorders) | 2 (2)
Inability to cannulate resulting in VWING removal (Blood and lymphatic system disorders) | 2 (2)
Sepsis (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venous Window Needle Guide (N=54)
Infiltration (Blood and lymphatic system disorders) | 13 (13)
Unable to cannulate (Blood and lymphatic system disorders) | 8 (8)
Stenosis (Blood and lymphatic system disorders) | 5 (5)
Infection (Infections and infestations) | 5 (5)
Thrombus (Blood and lymphatic system disorders) | 2 (2)
Seroma (Blood and lymphatic system disorders) | 2 (2)
Bruising (Blood and lymphatic system disorders) | 2 (2)
Pain (Blood and lymphatic system disorders) | 3 (3)
Possible dislodge VWING (Blood and lymphatic system disorders) | 1 (1)
Edema (Blood and lymphatic system disorders) | 1 (1)
Bleeding following cannulation (Blood and lymphatic system disorders) | 1 (1)
Incision dehiscence (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No